CLINICAL TRIAL: NCT05876637
Title: Effects of Left Nostril Breathing in Young Females Having Cardiovascular Hyper Reactivity to Cold Pressor Test.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Muqaddas Bibi
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: blood pressure; cold pressor test; heart rate
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Nostril Breathing (Experimental): The intervention protocol include healthy young females age 18-25 years.. All baseline measurements will be taken , Afterwards, the Cold pressor test would be performed for 1 minutes to induce acute stress while the BP would be monitored for every 30 seconds. At the end of the test, again the BP would be monitored. Out of all the recordings, the BP measuring the highest value would be recorded as final. We will then subtract the normal resting BP by highest value of the recording for each participant. Change in BP of systolic by 25mmHg and diastolic by 20mmHg will be considered hyper reactive. Then the hyper reactive subjects will be divided into two groups. Experimental group will receive left nostril breathing. CPT will be performed again at 4, 8 and 12 weeks to monitor the BP, heart rate and Spo2 likewise to check for any decline in sympathetic activity.
  Interventions: Other: Left Nostril Breathing
- Conventional (Active Comparator): The conventional protocol include healthy young females age 18-25 years. All baseline measurements will be taken, Afterwards, the Cold pressor test would be performed for 1 minutes to induce acute stress while the BP would be monitored for every 30 seconds. At the end of the test, again the BP would be monitored. Out of all the recordings, the BP measuring the highest value would be recorded as final. We will then subtract the normal resting BP by highest value of the recording for each participant. Change in BP of systolic by 25mmHg and diastolic by 20mmHg will be considered hyper reactive. Then the hyper reactive subjects will be divided into two groups Group A(Experimental) and Group B(Conventional). Controlled group will receive simple deep breathing exercises ,3 sessions per week for 12 weeks. CPT will be performed again at 4, 8 and 12 weeks to monitor the BP, heart rate and Spo2 likewise to check for any decline in sympathetic activity.
  Interventions: Other: Conventional

INTERVENTIONS:
Other: Left Nostril Breathing — The participants which will show cardiovascular hyper reactivity towards CPT will be divided into 2 groups having 30 participants in each group. Experimental group will receive Left Nostril Breathing(slow, deep breath taken through your left nostril while closing your right nostril with your right thumb. Then just as gently exhale long, slowly, and completely through the left nostril, just as gently. It will be done while sitting) for 10 minutes twice a day for the duration of 12 weeks. Follow up will be taken through administration Cold pressor test after every 4,8 and 12 weeks.
  Arms: Left Nostril Breathing
Other: Conventional — 30 participants will be recruited in conventional group which will receive simple deep breathing exercises of 3 sessions per week for the duration of 12 weeks.Follow up will be taken after every 4,8 and 12 weeks.
  Arms: Conventional

SUMMARY:
The purpose of this study is to evaluate the effects of left nostril breathing in young females having cardiovascular hyper reactivity to cold pressor test.Although,limited literature exist regarding hyper reactivity towards stress induced test in our youth and its effective and easy treatment in the form of left nostril breathing which could proves to be beneficial for our youth.

DETAILED DESCRIPTION:
The Cold Pressor Test (CPT) was introduced as a standard incentive for studying the vasomotor response (Hines and Brown 1932). Hyper-reactors were the subjects in his study who responded more strongly to CPT, Participants who show hyper reactivity to Cold pressor test (i.e. subjects showing 25 mmHg increase in systolic blood pressure along with 20 mmHg increase in diastolic blood pressure).They proposed that these hyper reactive could be candidates for hypertension in the future. Increased occurrence of these diseases could be attributed to an asymmetry in sympathetic and parasympathetic stimulation. Control or adaptation of breathing or breathing workouts i-e yoga are thought to be beneficial in the treatment of such disease. Although Yoga techniques proven to be effective in treating stress related disorders but it is time consuming and young population because of their busy routine couldn't be able to take out time for their health related issues. This study introduces very simple exercise in the form of left nostril breathing which decreases sympathetic activity and increases parasympathetic activity. It is inversely proportional to stress induced response of the body, it is very easy to perform and can be done at any time, and if found significantly effective for stress disorder ,it could be used in daily routine by our youth to get themselves prevented from major risk factors of CVD's particularly hypertension. This study will identify participants with a high potential risk of developing hypertension in the future by administering Cold pressor test, additionally the effects of left nostril breathing intervention on hyper reactive participants would be observed and if found significant, it would be a major breakthrough in primary prevention of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in the following category would be recruited into the study:
* Females Age (18-25) years
* Participants who show hyper reactivity to Cold pressor test (i.e subjects showing 25mmHg increase in systolic blood pressure along with 20mmHg increase in diastolic blood pressure)
* Consenting participants.

Exclusion Criteria:

* The participants in the following category would be excluded from the study:
* Participants on antihypertensive drugs.
* Participants who are diagnosed with any cardiovascular, renal, hepatic or metabolic disease.
* Participants having malignant tumor.
* Participants with nasal blockages, polyps ,Raynaud phenomena
* Females during menstrual cycle, pregnancy or on oral contraceptives.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Cold pressor test | After 4 weeks
  Cold pressor test will be conducted on participants to measure cardio vascular hyper reactivity to stress induce test.
Blood pressure | After 4 weeks
  Mercury sphygmomanometer will be used to measure blood pressure of participants
Heart Rate | After 4 weeks
  Pulse oximeter will be applied to the participant to measure their Heart rate.

SECONDARY OUTCOMES:
Oxygen saturation | after 4 weeks
  Pulse oximeter will be used on participant to measure Spo2.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Women Instritute of Rehabilitation Sciences, Jinnah College of Nursing, Abbottābād, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah N, Shah Q, Shah AJ. The burden and high prevalence of hypertension in Pakistani adolescents: a meta-analysis of the published studies. Arch Public Health. 2018 Apr 2;76:20. doi: 10.1186/s13690-018-0265-5. eCollection 2018. PMID 29619218
- [Background] Malhotra V, Srivastava R, Parasuraman P, Javed D, Wakode S, Thakare A, Sampath A, Kumari A. Immediate autonomic changes during right nostril breathing and left nostril breathing in regular yoga practitioners. J Educ Health Promot. 2022 Aug 25;11:280. doi: 10.4103/jehp.jehp_343_22. eCollection 2022. PMID 36325230
- [Background] Jain N, Srivastava RD, Singhal A. The effects of right and left nostril breathing on cardiorespiratory and autonomic parameters. Indian J Physiol Pharmacol. 2005 Oct-Dec;49(4):469-74. PMID 16579402
- [Background] Bargal S, Nalgirkar V, Patil A, Langade D. Evaluation of the Effect of Left Nostril Breathing on Cardiorespiratory Parameters and Reaction Time in Young Healthy Individuals. Cureus. 2022 Feb 18;14(2):e22351. doi: 10.7759/cureus.22351. eCollection 2022 Feb. PMID 35371755
- [Background] Wood DL, Sheps SG, Elveback LR, Schirger A. Cold pressor test as a predictor of hypertension. Hypertension. 1984 May-Jun;6(3):301-6. doi: 10.1161/01.hyp.6.3.301. PMID 6735451